CLINICAL TRIAL: NCT01859078
Title: Effect of Baricitinib on the Pharmacokinetics of Digoxin in Healthy Subjects
Brief Title: A Drug Drug Interaction (DDI) Study of Baricitinib (LY3009104) and Digoxin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14609; I4V-MC-JAGL (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — baricitinib; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Baricitinib + Digoxin (Experimental): Digoxin - 0.5 milligrams (mg) administered orally, twice daily (BID), 12 hours apart on Day 1. Then, 0.25 mg administered orally, once daily (QD) on Days 2 through 16.
  Baricitinib - 10 mg administered orally, QD, on Days 8 through 16.
  Interventions: Drug: Baricitinib; Drug: Digoxin

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104
Drug: Digoxin — Administered orally

SUMMARY:
The purpose of this study is to determine the effect of baricitinib on the levels of digoxin in the blood stream and how long it takes the body to remove digoxin. This study will also look at how safe and well-tolerated baricitinib is when given at the same time as digoxin in healthy participants. This study will last approximately 3-4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination
* Women not of child-bearing potential
* Menopausal women
* Have a body mass index of 18.0 to 29.0 kilograms per square meter (kg/m^2)

Exclusion Criteria:

* Women who are lactating
* Have previously completed or withdrawn from this study or any other study investigating baricitinib
* Currently enrolled in, have completed or discontinued within the last 90 days from a clinical trial involving an investigational product
* Have a pulse rate less than 50 beats per minute (bpm) at screening
* Have a current or recent history (less than 30 days prior to screening and/or less than 45 days prior to Day -1) of a clinically significant bacterial, fungal, parasitic, viral (not including rhinopharyngitis), or mycobacterial infection
* Have an absolute neutrophil count less than 2000 cells/microliter (2×10^9/liter) at screening or Day -1
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Have been exposed to a live vaccine within 12 weeks prior to the first dose or expected to need/receive a live vaccine
* Intend to use over-the-counter or prescription medication and/or herbal supplements within 14 days prior to dosing and during the study
* Have used or intend to use any drugs or substances that are known to be substrates, inducers, or inhibitors of P-glycoprotein (P-gp) within 30 days prior to dosing and throughout the study
* Have had symptomatic herpes zoster or herpes simplex infection within 90 days prior to the first dose

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri, 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leeds, West Yorkshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Baricitinib + Digoxin: Digoxin - 0.5 milligrams (mg) administered orally, twice daily (BID), 12 hours apart on Day 1. Then, 0.25 mg administered orally, once daily (QD) on Days 2 through 16.
  Baricitinib - 10 mg administered orally, QD, immediately prior to digoxin on Days 8 through 16.
Period: Overall Study
Arm/Group | Baricitinib + Digoxin
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Baricitinib + Digoxin: Digoxin - 0.5 mg administered orally, BID, 12 hours apart on Day 1. Then, 0.25 mg administered orally, QD on Days 2 through 16.
  Baricitinib - 10 mg administered orally, QD, immediately prior to digoxin on Days 8 through 16.
Arm/Group | Baricitinib + Digoxin
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 28

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve During 1 Dosing Interval (AUCτ) of Digoxin
Time Frame: Predose up to 24 hours post-dose on Days 7 and 16
Population: All enrolled participants who received study drug and had PK data to calculate AUCτ. Participants were analyzed based on the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*h/mL)
Groups:
- Digoxin Only: 0.5 mg digoxin administered orally, BID, 12 hours apart on Day 1. Then, 0.25 mg administered orally, QD on Days 2 through 7.
- Baricitinib + Digoxin: 10 mg baricitinib administered orally, QD, immediately prior to 0.25 mg digoxin administered orally, QD on Days 8 through 16.
Arm/Group | Digoxin Only | Baricitinib + Digoxin
Number analyzed (Participants) | 28 | 28
nanograms*hour/milliliter (ng*h/mL) | 18.7 (18) | 16.8 (20)

2. Primary Outcome: PK: Maximum Concentration (Cmax) of Digoxin
Time Frame: Predose up to 24 hours post-dose on Days 7 and 16
Population: All enrolled participants who received study drug and had PK data to calculate Cmax. Participants were analyzed based on the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Digoxin Only | Baricitinib + Digoxin
Number analyzed (Participants) | 28 | 28
nanograms/milliliter (ng/mL) | 2.04 (23) | 1.80 (20)

3. Primary Outcome: PK: Time of Maximum Observed Drug Concentration (Tmax) of Digoxin
Time Frame: Predose up to 24 hours post-dose on Days 7 and 16
Population: All enrolled participants who received study drug and had PK data to calculate tmax. Participants were analyzed based on the treatment they received.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Digoxin Only | Baricitinib + Digoxin
Number analyzed (Participants) | 28 | 28
hours (h) | 1.00 [0.50 to 2.00] | 1.00 [0.42 to 2.00]

4. Secondary Outcome: PK: Amount of Drug Excreted Unchanged During 1 Dosing Interval (Aeτ) of Digoxin
Time Frame: 0 to 24 hours post-dose on Days 7 and 16
Population: All enrolled participants who received study drug and had PK data to calculate Aeτ. Participants were analyzed based on the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams (mg)
Arm/Group | Digoxin Only | Baricitinib + Digoxin
Number analyzed (Participants) | 28 | 28
milligrams (mg) | 0.177 (18) | 0.155 (22)

5. Secondary Outcome: PK: Renal Clearance (CLr) of Digoxin
Description: CLr is the volume of plasma from which study drug is completely removed by the kidney in a given time and is calculated as Aeτ divided by AUCτ.
Time Frame: Predose to 24 hours post-dose on Days 7 and 16
Population: All enrolled participants who received study drug and had PK data to calculate CLr. Participants were analyzed based on the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour (L/h)
Arm/Group | Digoxin Only | Baricitinib + Digoxin
Number analyzed (Participants) | 28 | 28
Liters/hour (L/h) | 9.46 (20) | 9.20 (18)

ADVERSE EVENTS:
Arm/Group | Digoxin Only | Baricitinib + Digoxin
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 10/28 | 6/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Digoxin Only (N=28) | Baricitinib + Digoxin (N=28)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Fatigue (General disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 2 (3)
Pollakiuria (Renal and urinary disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days